CLINICAL TRIAL: NCT01204762
Title: Dose-Ranging Study to Evaluate the Safety, Efficacy and Pharmacokinetics of Pegylated Interferon Lambda (BMS-914143) Monotherapy in Interferon-Naive Patients With Chronic Hepatitis B Virus Infection Who Are HBeAg-positive
Brief Title: Dose Ranging Study of Pegylated Interferon Lambda in Patients With Hepatitis B and Positive for the Hepatitis B e Antigen
Acronym: LIRA-B
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AI452-005; 2010-020387-38 (EudraCT Number)
Record Dates: First submitted 2010-09-16; First posted 2010-09-17 (Estimated); Last update posted 2015-10-09 (Estimated); Status verified 2015-09

CONDITIONS: Hepatitis B Virus
MeSH Terms: conditions — Hepatitis B | interventions — peginterferon alfa-2a; peginterferon lambda-1a; entecavir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Part A Arm 1: pegIFN (180 μg) (Experimental)
  Interventions: Drug: pegIFN
- Part A Arm 2: pegIFNα-2a (Active Comparator)
  Interventions: Drug: pegIFNα-2a
- Part B: pegIFN lambda + Entecavir (Experimental)
  Interventions: Drug: PegIFN lambda; Drug: Entecavir

INTERVENTIONS:
Drug: pegIFN — Syringe, Subcutaneous, 180 μg, Once Weekly, 48 weeks
  Arms: Part A Arm 1: pegIFN (180 μg)
Drug: pegIFNα-2a — Syringe, Subcutaneous 180 μg, Once Weekly, 48 Weeks
  Other Names: Pegasys
  Arms: Part A Arm 2: pegIFNα-2a
Drug: PegIFN lambda — Syringe, Subcutaneous, 180 µg, Once weekly, 48 weeks
  Other Names: BMS-914143
  Arms: Part B: pegIFN lambda + Entecavir
Drug: Entecavir — Tablet, Oral, 0.5 mg, Once daily, 12 weeks initial monotherapy followed by 48 weeks of combination therapy with PegIFN lambda
  Other Names: Baraclude
  Arms: Part B: pegIFN lambda + Entecavir

SUMMARY:
At least 1 dose of pegIFNλ will be identified which is safe, well tolerated, and efficacious for the treatment of chronic hepatitis B virus infection (CHB)

Amendment 7, Part B Sub Study: The primary purpose of this amendment is to obtain preliminary data on the safety of pegylated interferon Lambda (Lambda) when administered in combination with Entecavir(ETV) to patients with hepatitis E antigen-positive (HBeAg-positive) chronic hepatitis B(CHB) infection employing a sequential therapy approach

DETAILED DESCRIPTION:
Part B sub study is Open Label

ELIGIBILITY:
Inclusion Criteria:

* Infection with the hepatitis B virus (HBV) and positive for the hepatitis B e antigen
* Between the ages of 18 and 70
* Have not been previously treated with an interferon
* HBV nucleos(t)ide-naive

Exclusion Criteria:

* Not infected with the hepatitis C virus (HCV), hepatitis D virus (HDV) or human immunodeficiency virus (HIV)
* Do not have a serious liver, psychiatric, blood, thyroid, lung, heart or eye disease
* Able to tolerate oral medication

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2010-11; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Part A: Proportion of subjects who achieve Hepatitis B e antigen (HBeAg) seroconversion | 24 weeks post-dosing (Week 72)
Part A: Number and percent of subjects with serious adverse events (SAEs) and discontinuations due to adverse events | Week 24
Part A: Number and percent of subjects with serious adverse events (SAEs) and discontinuations due to adverse events | 24 weeks post-dosing (Week 72)
Part B: Safety and tolerability of Lambda/ETV regimen as measured by the frequency of SAEs and discontinuations due to AEs | Up to 84 Weeks

SECONDARY OUTCOMES:
Part A: Proportion of subjects who achieve an hepatitis B virus Deoxyribonucleic acid levels (HBV DNA) < 50 IU/mL (approximately 300 copies/mL) using the Roche COBAS® TaqMan - High Pure System (HPS) assay | Weeks 24, 48, 72, 96, 120, 144, 168 and 192
Part A: Mean change from baseline in log10 HBV DNA levels over time (Proportion of subjects with Alanine amino transferase (ALT) normalization (≤ 1 x upper limit of normal (ULN)) | Baseline (Day 1), Weeks 24, 48, 72, 96, 120, 144, 168 and 192
Part A: Proportion of subjects with ALT normalization (≤ 1 x ULN) | Weeks 24, 48, 72, 96, 120, 144, 168 and 192
Part A: Hepatitis E antigen (HBeAg) loss | Weeks 24, 48, 72, 96, 120, 144, 168 and 192
Part A: HBeAg seroconversion | Weeks 24, 48, 96, 120, 144, 168 and 192
Part A: Mean change from baseline in log10 quantitative HBeAg levels over time | Baseline (Day 1), Weeks 24, 48, 96, 120, 144, 168 and 192
Part A: Number and percent of subjects with adverse events (AEs) or laboratory abnormalities | Up to Week 24
Part A: Number and percent of subjects with adverse events (AEs) or laboratory abnormalities | Up to Week 72
Part A: Pharmacokinetic (PK) parameter Maximum observed concentration (Cmax) of Pegylated interferon lambda (pegIFNλ) will be derived from serum concentration versus time data | Day 1 (including intense PK), Weeks 2, 4, 12 (including intense PK), 16, 24, 40, 48
Part A: Pharmacokinetic (PK) parameter Time of maximum observed concentration (Tmax) of Pegylated interferon lambda (pegIFNλ) will be derived from serum concentration versus time data | Day 1 (including intense PK), Weeks 2, 4, 12 (including intense PK), 16, 24, 40, 48
Part A: Pharmacokinetic (PK) parameter Trough serum concentration pre-dose (C0) of Pegylated interferon lambda (pegIFNλ) will be derived from serum concentration versus time data | Day 1 (including intense PK), Weeks 2, 4, 12 (including intense PK), 16, 24, 40, 48
Part A: PK parameter serum concentration 168 hours post observed dose [Cmin] (C0 will be used as an estimate of Cmin if sample is not collected) of pegIFNλ will be derived from serum concentration versus time data | Day 1 (including intense PK), Weeks 2, 4, 12 (including intense PK), 16, 24, 40, 48
Part A: PK parameter Area under the concentration-time curve in 1 dosing interval from time 0 to 168 hours post observed dose [AUC(TAU)] of pegIFNλ will be derived from serum concentration versus time data | Day 1 (including intense PK), Weeks 2, 4, 12 (including intense PK), 16, 24, 40, 48
Part A: PK parameter Accumulation index (AI) ratio of AUC(TAU) at steady-state to AUC(TAU) after the first dose (only conducted if data warrant) of pegIFNλ will be derived from serum concentration versus time data | Day 1 (including intense PK), Weeks 2, 4, 12 (including intense PK), 16, 24, 40, 48
Part B: HBeAg seroconversion rate at 24 weeks off treatment | Week 84
Part B: Antiviral activity of Lambda/ETV regimen, as determined by the proportion of subjects who achieve an HBV DNA < 50 IU/mL (approximately 300 copies/mL) using the Roche COBAS® TaqMan - HPS assay | Weeks 4, 8, 12, 24, 36, 60, and 84
Part B: Mean change from baseline in HBV DNA over time in subjects treated with Lambda/ETV | Weeks 4, 8, 12, 24, 36, 60, and 84
Part B: HBeAg loss and seroconversion in subjects treated with Lambda/ETV regimen | Weeks 12, 24, 36, 60 and 84
Part B: HBeAg levels over time in subjects treated with Lambda/ETV regimen | Weeks 4, 8, 12, 24, 36, 60, and 84
Part B: biochemical response rates in subjects treated with Lambda/ETV regimen | Weeks 4, 8, 12, 24, 36, 60, and 84
Part B: Pharmacokinetic (PK) parameter Maximum observed concentration (Cmax) of Lambda/ETV regimen will be derived from serum concentration versus time data | Baseline (Day 1), Weeks 4, 12, 16, 24, 52, 60
Part B: Pharmacokinetic (PK) parameter Time of maximum observed concentration (Tmax) of Lambda/ETV regimen will be derived from serum concentration versus time data | Baseline (Day 1), Weeks 4, 12, 16, 24, 52, 60
Part B: Pharmacokinetic (PK) parameter Trough serum concentration pre-dose (C0) of Lambda/ETV regimen will be derived from serum concentration versus time data | Baseline (Day 1), Weeks 4, 12, 16, 24, 52, 60
Part B: PK parameter Area under the concentration-time curve in 1 dosing interval from time 0 to 168 hours post observed dose [AUC(TAU)] of Lambda/ETV regimen will be derived from serum concentration versus time data | Baseline (Day 1), Weeks 4, 12, 16, 24, 52, 60
Part B: PK parameter serum concentration 168 hours post observed dose [Cmin] (C0 will be used as an estimate of Cmin if sample is not collected) of Lambda/ETV regimen will be derived from serum concentration versus time data | Baseline (Day 1), Weeks 4, 12, 16, 24, 52, 60
Part B: PK parameter Accumulation index (AI) ratio of AUC(TAU) at steady-state to AUC(TAU) after the first dose (only conducted if data warrant) of Lambda/ETV regimen will be derived from serum concentration versus time data | Baseline (Day 1), Weeks 4, 12, 16, 24, 52, 60
Part B: Rate of resistance to ETV during treatment with the Lambda/ETV regimen | Up to Week 84

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (48):
- United States (13):
  - Advanced Clinical Research Institute, Anaheim, California
  - Sc Clinical Research, Inc., Garden Grove, California
  - University Of California, Davis Medical Center, Sacramento, California
  - Research And Education, Inc., San Diego, California
  - Yale New Haven Hospital, New Haven, Connecticut
  - Atlanta Gastroenterology Associates, Llc, Atlanta, Georgia
  - Mercy Medical Center, Baltimore, Maryland
  - Gastro Center Of Maryland, Colombia, Maryland
  - Medical Procare, Pllc, Flushing, New York
  - Office Of Sing Chan Md, Flushing, New York
  - Duke University Medical Center, Durham, North Carolina
  - Oregon Health & Science University, Portland, Oregon
  - University Of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
- Australia (7):
  - Local Institution, Camperdown, New South Wales
  - Local Institution, Liverpool, New South Wales
  - Local Institution, Westmead Nsw, New South Wales
  - Local Institution, Clayton Vic, Victoria
  - Local Institution, Heidelberg Vic, Victoria
  - Local Institution, Melbourne, Victoria
  - Local Institution, Fremantle, Western Australia
- Canada (4):
  - Heritage Medical Research Clinic, University Of Calgary, Calgary, Alberta
  - Local Institution, Winnipeg, Manitoba
  - Toronto General Hospital, Toronto, Ontario
  - Toronto Western Hospital University Health Network, Toronto, Ontario
- France (4):
  - Local Institution, Clichy
  - Local Institution, Nice
  - Local Institution, Paris
  - Local Institution, Rennes
- Germany (5):
  - Local Institution, Frankfurt
  - Local Institution, Freiburg im Breisgau
  - Local Institution, Hamburg
  - Local Institution, Hanover
  - Local Institution, Tübingen
- Hong Kong (3):
  - Local Institution, Hong Kong
  - Local Institution, Shatin
  - Local Institution, Tai Po
- Italy (2):
  - Local Institution, Florence
  - Local Institution, Roma
- Local Institution, Rotterdam, Netherlands
- Local Institution, Singapore, Singapore
- South Korea (3):
  - Local Institution, Chuncheon
  - Local Institution, Gyeonggi-do
  - Local Institution, Seoul
- Taiwan (5):
  - Local Institution, Kaohsiung City
  - Local Institution, Taichung
  - Local Institution, Tainan
  - Local Institution, Taipei
  - Local Institution, Taoyuan District

REFERENCES:
- [Derived] Phillips S, Mistry S, Riva A, Cooksley H, Hadzhiolova-Lebeau T, Plavova S, Katzarov K, Simonova M, Zeuzem S, Woffendin C, Chen PJ, Peng CY, Chang TT, Lueth S, De Knegt R, Choi MS, Wedemeyer H, Dao M, Kim CW, Chu HC, Wind-Rotolo M, Williams R, Cooney E, Chokshi S. Peg-Interferon Lambda Treatment Induces Robust Innate and Adaptive Immunity in Chronic Hepatitis B Patients. Front Immunol. 2017 May 29;8:621. doi: 10.3389/fimmu.2017.00621. eCollection 2017. PMID 28611778
- [Derived] Chan HLY, Ahn SH, Chang TT, Peng CY, Wong D, Coffin CS, Lim SG, Chen PJ, Janssen HLA, Marcellin P, Serfaty L, Zeuzem S, Cohen D, Critelli L, Xu D, Wind-Rotolo M, Cooney E; LIRA-B Study Team. Peginterferon lambda for the treatment of HBeAg-positive chronic hepatitis B: A randomized phase 2b study (LIRA-B). J Hepatol. 2016 May;64(5):1011-1019. doi: 10.1016/j.jhep.2015.12.018. Epub 2015 Dec 29. PMID 26739688
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx